CLINICAL TRIAL: NCT06168578
Title: The Effect of Alveolar Recruitment Manoeuvre on Optic Nerve Sheath Diameter in Laparoscopic Hysterectomies
Status: Active, not recruiting | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Nazan KOCAOGLU, MD, assistant professor, Balikesir University
Other Study IDs: ARM-ONSD-22-01
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Recruitment; Optic Nerve; Hysterectomy
Keywords: alveolar recruitment; optical diameter; laparoscopic hysterectomy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I (ARM-): After intubation, 5 cmH2O PEEP will be applied until the end of the operation: * First ONSD measurement will be performed 5 minutes after intubation with the patient in supine position (T0)
  * A second ONSD measurement will be performed 10 minutes after intubation with the patient in supine position. (T1)
  * ONSD will be measured for the third time 5 minutes after pneumoperitoneum is established with 12-13 mmHg. (T2)
  * At 10 minutes of Trendelenburg position (45⁰), ONSD will be measured for the fourth time (T3).
  * In Trendelenburg position (45⁰), ONSD will be measured for the fifth time after removal of the uterus. (T4)
  * After the supine position is assumed before extubation and pneumoperitoneum is terminated, ONSD will be measured for the sixth time before the neuromuscular blocker is reversed. (T5)
  Interventions: Device: ultrasound
- Group II (ARM+): After intubation, 5 cmH2O PEEP will be applied until the end of the operation: * ONSD will be measured 5 minutes after intubation with the patient in supine position (T0)
  * ARM will be applied 10 minutes after intubation, and ONSD will be measured for the second time when the peak pressure is reached. (T1)
  * ONSD will be measured for the third time 5 minutes after pneumoperitoneum is established with 12-13 mmHg. (T2)
  * At 10 minutes of Trendelenburg position (45⁰), ONSD will be measured for the fourth time (T3).
  * Trendelenburg position (45⁰), ARM will be applied after the uterus is removed, and ONSD will be measured for the fifth time when the peak pressure is reached. (T4)
  * After the supine position is assumed before extubation and pneumoperitoneum is terminated, ONSD will be measured for the sixth time before the neuromuscular blocker is reversed. (T5)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Optic nerve diameter will be measured by ultrasound at certain stages of the operation in Group I (ARM-) and Group II (ARM+)

SUMMARY:
Laparoscopic total hysterectomy is the most common gynaecological surgical procedure after caesarean section. In laparoscopic total hysterectomy, intraabdominal pressure increases, venous return decreases, hypercarbia and acidosis may occur due to pneumoperitoneum due to CO2 insufflation and upright trendelenburg position (TP). Cerebral blood flow, intracranial pressure (ICP) and intraocular pressure (IOP) increase. One study showed that TP and an intraabdominal pressure of mmHg significantly increased ICP.

CO2 insufflation into the abdominal cavity causes upward displacement of the diaphragm, resulting in an increased risk of regurgitation, decreased lung volumes and compliance, atelectasis, increased airway resistance and ventilation-perfusion mismatch. At the same time, combined with the effects of general anaesthesia, a decrease in partial arterial oxygen pressure (PaO2) is expected in patients. The alveolar recirculation manoeuvre (ARM), is based on the technique of opening atelectatic lung fields by keeping the airway pressure high for a while. This manoeuvre can be performed with methods such as PEEP, CPAP, and pressure-controlled mechanical ventilation. High PEEP application may cause an increase in ICP and a decrease in cerebral perfusion pressure by increasing intrathoracic pressure and decreasing cerebral venous return. Therefore, intracranial pressure monitoring should be performed especially in patients with PEEP above 8-10 cmH2O.

Intraventricular and intraparenchymal measurements, which are the gold standard methods for ICP monitoring, are invasive procedures with various risks. Noninvasive methods such as cranial CT, brain MRI, transcranial Doppler, and measurement of optic nerve sheath diameter (ONSD) can also be used for ICP measurement. Ultrasonography of the optic nerve sheath diameter is an increasingly common method because it is noninvasive and can be performed at the bedside. The optic nerve sheath is the continuation of the transverse subarachnoid space and the cerebral duramater. It is connected to the intracranial subarachnoid space with cerebrospinal fluid. Therefore, an increase in ICP increases the optic nerve sheath diameter (ONSD). Maissan et al. They think that ONSD reflects the changes in ICP simultaneously. The aim of this study was to evaluate the effect of ARM on intracranial pressure in patients undergoing total laparoscopic hysterectomy under general anaesthesia using optic nerve sheath diameter.

DETAILED DESCRIPTION:
METHODS AND MATERIALS

Inclusion Criteria:

* Elective total laparoscopic hysterectomy under general anaesthesia
* 18-65 years
* ASA I-II
* Female volunteers with a body mass index (BMI) ≤35 kg/m2 with written informed consent will be included in the study

Exclusion Criteria:

* Previous eye surgery, ophthalmic disease
* Previous neurosurgery
* Transient ischaemic attack, other neurological diseases affecting the eye or that may affect ICP
* Previous lung surgery, pneumothorax
* Pulmonary diseases (emphysema, pneumonia, malignancy)
* Patients in whom the surgical plan has changed (open/complicated surgery) will not be included in the study

Anaesthesia Administration:

All volunteers who will participate in the study will be informed, written informed consent will be obtained and demographic data will be recorded. After providing a preoperative 20 G intravenous (IV) line, 10 mL/kg/hour balanced crystalloid fluid infusion will be started. All volunteers will undergo standard monitoring (ECG, heart rate, non-invasive blood pressure, SPO2, temperature) and neuromuscular monitoring (Train of four). These parameters will be recorded at 5 minute intervals and simultaneously with ONSD measurement times (T0-T5) until the end of the operation in both groups. Anaesthesia induction will be provided with 2 mg/kg propofol (Propofol-Pf 1%, 200 mg/20 mL- Polifarma) and 1 μg/kg fentanyl (Fentaver 0.5 mg/10 mL-Haver Farma) IV as standard. For muscle relaxation, 0.6 mg/kg rocuronium (Muscobloc 50 mg/5 mL-Polifarma) will be administered IV. When the train of four rate (TOFR) response is zero, the patient will be intubated orotracheally. (During the operation, if a neuromuscular blocker is needed according to TOFR, IV 0.1 mg/kg rocuronium will be administered additionally) After intubation, gastric decompression will be provided by applying an orogastric tube. Anaesthesia maintenance will be performed with 0.5 L/min fresh gas flow, tidal volume 6-8 mL/kg, oxygen concentration with inspiratory oxygen level between 40-45, sevoflurane (Sevorane-AbbVie) with minimum alveolar concentration (MAK) 0.9-1.1. Mechanical ventilation will be performed with Volume Auto Flow mode (V-AF) with ETCO2 between 35-45 mmHg.

After intubation, volunteers will be divided into 2 groups according to a computerised randomisation scheme by an anaesthetist not involved in the study. During the operation, follow-up of the volunteers and ARM application will be performed by the same anaesthetist, and ONSD measurement will be performed by another experienced anaesthesiologist.

Group I (ARM-): 5 cmH2O PEEP will be applied after intubation until the end of the operation

* First ONSD measurement will be performed 5 minutes after intubation with the patient in supine position (T0)
* A second ONSD measurement will be performed 10 minutes after intubation with the patient in supine position. (T1)
* ONSD will be measured for the third time 5 minutes after pneumoperitoneum is established with 12-13 mmHg. (T2)
* At 10 minutes of Trendelenburg position (45⁰), ONSD will be measured for the fourth time (T3).
* In Trendelenburg position (45⁰), ONSD will be measured for the fifth time after removal of the uterus. (T4)
* After the supine position is assumed before extubation and pneumoperitoneum is terminated, ONSD will be measured for the sixth time before the neuromuscular blocker is reversed. (T5)

Group II (ARM+): After intubation, 5 cmH2O PEEP will be applied until the end of the operation

* ONSD will be measured 5 minutes after intubation with the patient in supine position. (T0)
* ARM will be applied 10 minutes after intubation, and ONSD will be measured for the second time when the peak pressure is reached. (T1)
* ONSD will be measured for the third time 5 minutes after pneumoperitoneum is established with 12-13 mmHg. (T2)
* At 10 minutes of Trendelenburg position (45⁰), ONSD will be measured for the fourth time (T3).
* Trendelenburg position (45⁰), ARM will be applied after the uterus is removed, and ONSD will be measured for the fifth time when the peak pressure is reached. (T4)
* After the supine position is assumed before extubation and pneumoperitoneum is terminated, ONSD will be measured for the sixth time before the neuromuscular blocker is reversed. (T5)

ARM application:

The alveolar recruitment manoeuvre (ARM) will be performed with the automatic recruitment application available in anaesthesia devices. ARM will be performed by gradually increasing PEEP and plateau pressure at a constant driving pressure of 12-15 cmH2O in pressure-controlled ventilation. PEEP will be increased from 5 cmH2O to 20 cmH2O. The plateau pressure will be increased to 40 cmH2O and 10 breaths will be performed at this level. After 10 consecutive breaths, the target PEEP will be gradually decreased from 20 cmH2O and kept constant at 5 cmH2O.

ONSD measurement:

ONSD of the patient volunteers included in the study will be measured by ultrasonographic method; a total of 6 times (T0, T1, T2, T3, T3, T4, T5), each time in both eyes. Water-soluble sterile thick gel layer will be applied to the closed upper eyelid and a linear 10-5 MHz (Sonosite M-Turbo) ultrasound probe will be gently placed. Carefully and without applying excessive pressure, the entrance of the optic nerve to the orbital globe will be visualised on the monitor in 2D mode. After finding the optimum contrast between the retrobulbar echogenic fatty tissue and the vertical hypoechogenic band, the diameter of the optic nerve sheath will be measured 3 mm behind the optic disc. The gel applied after the measurement will be wiped off with a clean napkin. ONSD measurements; transverse measurements of both eyes will be made three times, averaged and recorded. ONSD measurements will be performed by an experienced anaesthetist who will be called to the operation room only during ONSD measurements.

The patient volunteers will undergo standard surgical procedure and will be operated in 45⁰ trendelenburg position with a pneumoperitoneum pressure of 12-13 mmHg. The time between CO2 insufflation and desufflation will be recorded as "pneumoperitoneum time". Hypotension will be defined as systolic arterial pressure decreases by 30% compared to baseline. In treatment, 250 mL 0.9% NaCl rapid infusion will be administered first. If no response is obtained, 10 mg ephedrine will be given IV. When bradycardia occurs (heart rate <50 beats/min), 0.5 mg atropine IV will be administered. The time from the skin incision until the end of the surgical procedure will be recorded as "operation time".

Sevoflurane flow will be terminated 15 minutes before the end of the operation. Patient volunteers will receive 100 mg tramadol HCl (Tradolex 100 mg/2 mL-Menta Pharma) IV and 1 g paracetamol (Partemol 1 g/ 100 mL- VEM pharmaceuticals) IV infusion. Fresh gas flow will be increased to 8 L/min at the end of the operation. For the termination of neuromuscular blockade, 4 mg/kg sugammadex (Brimadeks 200 mg/ 2 mL-Polifarma) will be administered IV. Volunteers will be extubated with a TOFR of 0.9 and transferred to the postoperative recovery unit (PACU). The time between induction of anaesthesia and extubation will be recorded as "anaesthesia time".

ELIGIBILITY:
Inclusion Criteria:

* Elective total laparoscopic hysterectomy under general anaesthesia
* 18-65 years
* ASA I-II
* Female volunteers with a body mass index (BMI) ≤35 kg/m2 with written informed consent will be included in the study

Exclusion Criteria:

* Previous eye surgery, ophthalmic disease
* Previous neurosurgery
* Transient ischaemic attack, other neurological diseases affecting the eye or that may affect ICP
* Previous lung surgery, pneumothorax
* Pulmonary diseases (emphysema, pneumonia, malignancy)
* Patients in whom the surgical plan has changed (open/complicated surgery) will not be included in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 18-65 years
  * Female volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
ICP | inoperation
  The aim of this study was to evaluate the effect of alveolar recruitment manoeuvre (ARM) on intracranial pressure in patients undergoing total laparoscopic hysterectomy under general anaesthesia using the diameter of the optic nerve sheath.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Kocaoglu, Principal Investigator — Balikesir University
Locations (1):
- Balikesir University Faculty of Medicine, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, it can be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: After the study is completed
Access Criteria: only university researchers

REFERENCES:
- [Background] Huynh T, Messer M, Sing RF, Miles W, Jacobs DG, Thomason MH. Positive end-expiratory pressure alters intracranial and cerebral perfusion pressure in severe traumatic brain injury. J Trauma. 2002 Sep;53(3):488-92; discussion 492-3. doi: 10.1097/00005373-200209000-00016. PMID 12352486
- [Background] Killer HE, Laeng HR, Flammer J, Groscurth P. Architecture of arachnoid trabeculae, pillars, and septa in the subarachnoid space of the human optic nerve: anatomy and clinical considerations. Br J Ophthalmol. 2003 Jun;87(6):777-81. doi: 10.1136/bjo.87.6.777. PMID 12770980
- [Background] Maissan IM, Dirven PJ, Haitsma IK, Hoeks SE, Gommers D, Stolker RJ. Ultrasonographic measured optic nerve sheath diameter as an accurate and quick monitor for changes in intracranial pressure. J Neurosurg. 2015 Sep;123(3):743-7. doi: 10.3171/2014.10.JNS141197. Epub 2015 May 8. PMID 25955869